CLINICAL TRIAL: NCT02000518
Title: Phase 1 Study of Neurological Outcome After Emergency Radiotherapy in Metastatic Spinal Cord Compression
Brief Title: Emergency Radiotherapy in Metastatic Spinal Cord Compression of Patients With Non-small Cell Lung Cancer
Acronym: CK-INF
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Alexandra Jensen, Neurological outcome after emergency radiotherapy in MSCC of patients with non-small cell lung cancer, Heidelberg University
Other Study IDs: S-514/2011
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Neurological Outcome; Survival From First Diagnosis Metastatic Spinal Cord Compression to Death
Keywords: emergency radiotherapy; MSCC; spine; neurological outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- external beam radiotherapy: emergency radiotherapy within 12 hours after neurological deficit due to MSCC
  Interventions: Radiation: external beam radiotherapy

INTERVENTIONS:
Radiation: external beam radiotherapy

SUMMARY:
Acute neurological deficit in metastatic spinal cord compression is an emergency condition in radiation oncology. Despite some reports about the high efficacy of radiation treatment for oncological emergencies, a standard of care is not well defined, especially the time interval of immediate RT after deficit, and neurological outcome with respect to poor survival in non-small cell lung cancer patients. The objective of this trial is to investigate neurological outcome after emergency radiotherapy in metastatic spinal cord compression of non-small cell lung cancer patients with acute neurological deficit.

DETAILED DESCRIPTION:
Subjects and recruitment 15 consecutive patients with histologically confirmed non-small cell lung cancer and bone metastases of the thoracic or lumbar segments of the vertebral column will be screened for this trial in the Radiooncology Department of the Heidelberg University Clinic. Inclusion criteria are an age of 18 to 80 years, acute neurological symptom caused by metastatic spinal cord compression, no radiotherapy in this spinal area before, and written consent to participate.

Design and procedures This is a prospective, controlled, explorative trial to investigate the neurological outcome after emergency radiotherapy in metastatic spinal cord compression of non-small cell lung cancer patients with acute neurological deficit. RT start within 12 hours after onset of neurological symptoms. The target parameters will be measured at the start of radiotherapy (t0), and six weeks after radiotherapy (RT) (t1). The target parameters comprise the documentation and completion of the ASIA Impairment Scale (AIS), and the recording of patient-specific data.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are an age of 18 to 80 years, acute neurological symptom caused by metastatic spinal cord compression, no RT in this spinal area before, and written consent to participate.

Exclusion Criteria:

* neurological symptom more than 12 hours before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: histologically confirmed non-small cell lung cancer and bone metastases of the thoracic or lumbar segments of the vertebral column
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
neurological outcome | 6 weeks after end of radiotherapy
  The primary endpoint was neurological outcome, assessed using the ASIA Impairment Scale (AIS)

SECONDARY OUTCOMES:
local control | 6 weeks after end of radiotherapy
  according CT scan, local control will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Heidelberg, Departement radiation oncology, Heidelberg, Germany

REFERENCES:
- [Background] Rades D, Fehlauer F, Schulte R, Veninga T, Stalpers LJ, Basic H, Bajrovic A, Hoskin PJ, Tribius S, Wildfang I, Rudat V, Engenhart-Cabilic R, Karstens JH, Alberti W, Dunst J, Schild SE. Prognostic factors for local control and survival after radiotherapy of metastatic spinal cord compression. J Clin Oncol. 2006 Jul 20;24(21):3388-93. doi: 10.1200/JCO.2005.05.0542. PMID 16849752
- [Background] Bach F, Larsen BH, Rohde K, Borgesen SE, Gjerris F, Boge-Rasmussen T, Agerlin N, Rasmusson B, Stjernholm P, Sorensen PS. Metastatic spinal cord compression. Occurrence, symptoms, clinical presentations and prognosis in 398 patients with spinal cord compression. Acta Neurochir (Wien). 1990;107(1-2):37-43. doi: 10.1007/BF01402610. PMID 2096606
- [Background] Christian E, Adamietz IA, Willich N, Schafer U, Micke O; German Working Group Palliative Radiotherapy; German Society for Radiation Oncology (DEGRO). Radiotherapy in oncological emergencies--final results of a patterns of care study in Germany, Austria and Switzerland. Acta Oncol. 2008;47(1):81-9. doi: 10.1080/02841860701481554. PMID 17851852
- [Derived] Rief H, Heinhold RC, Petersen LC, Rieken S, Bruckner T, Moghaddam-Alvandi A, Debus J, Sterzing F. Neurological outcome after emergency radiotherapy in MSCC of patients with non-small cell lung cancer--a prospective trial. Radiat Oncol. 2013 Dec 28;8:297. doi: 10.1186/1748-717X-8-297. PMID 24373638